CLINICAL TRIAL: NCT07323082
Title: Role of Purinergic Compounds in the Vascular Pathology of Pseudoxanthoma Elasticum
Brief Title: Purinergic Compounds in Pseudoxanthoma Elasticum
Acronym: PURI-PXE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nice (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 25-PP-14
Record Dates: First submitted 2025-12-16; First posted 2026-01-07 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-12

CONDITIONS: Pseudoxanthoma Elasticum
Keywords: ppi; ADO; vascular pathology
MeSH Terms: conditions — Pseudoxanthoma Elasticum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PXE Patient (Experimental): PXE Patient
  Interventions: Biological: supplementary tubes
- NON PXE Patient (Other): NON PXE Patient
  Interventions: Biological: supplementary tubes; Radiation: SCANNER

INTERVENTIONS:
Biological: supplementary tubes — * One 2.5 ml EDTA blood tube for PPi measurement.
  * Special blotting paper for collecting blood drops for ADO measurement.
  * 7.5 ml whole blood for ectoenzyme measurement
Radiation: SCANNER — non-injected coronary and lower limb scanner
  Arms: NON PXE Patient

SUMMARY:
Pseudoxanthoma elasticum (PXE) is a rare genetic disorder, transmitted as an autosomal recessive trait, affecting approximately 1 in 50,000 people, predominantly women. It is characterised by progressive calcification of tissues rich in elastic fibres, particularly the skin, retina and arteries. It often begins in young adults and can eventually lead to central blindness, peripheral artery disease, strokes, tendon pain, recurrent kidney stones and visible skin changes.

The diagnosis is based on clinical examination (skin papules, angioid streaks) and can be confirmed by biopsy or genotyping of the ABCC6 gene, whose mutation leads to extracellular ATP deficiency. This deficiency reduces the production of pyrophosphate (PPi), a natural inhibitor of calcification, thus promoting abnormal calcium deposits in tissues. To date, there is no curative treatment, but clinical trials are evaluating oral administration of PPi, with encouraging results.

The role of purinergic metabolism is increasingly being explored in PXE. The cascade of conversion of ATP to adenosine (ADO) via ectonucleotidase pyrophosphatase 1 (ENPP1) and 5' ectonucleotidase (NT5E) indirectly regulates the activity of tissue-nonspecific alkaline phosphatase (TNAP), an enzyme that degrades PPi. An imbalance in this cascade could aggravate calcifications. The joint measurement of PPi, ADO and these enzymes, which has recently become possible, could not only refine our understanding of the disease, but also pave the way for new therapeutic strategies.

ELIGIBILITY:
Inclusion Criteria:

* Male or female,
* Age >18 years
* Covered by social security,
* Informed and having signed the informed consent form.

PXE patients:

- with PXE defined according to current clinical criteria for PXE (REACT-PXE and PNDS consensus) and with an ABCC6 mutation.

Exclusion Criteria:

* Patients treated with bisphosphonates, vitamin K antagonists, and dietary supplements containing calcium, phosphates, magnesium, zinc, or iron.
* Treatments likely to alter adenosine levels (caffeine, salbutamol, beta-blockers, etc.).
* Progressive bone diseases (osteoporosis, chondrocalcinosis, gout, etc.).
* Progressive and/or treated cancerous diseases.
* Progressive and/or treated inflammatory or autoimmune diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2026-01-15 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
potential role of the ADO | at inclusion
  mesure of concentration

SECONDARY OUTCOMES:
correlation between ADO, PPi and ectoenzymatic activities | at inclusion
  correlation between concentrations
correlation between ADO, PPi and calcification score | at inclusion
  correlation between concentrations and calcification score (%)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Angers University hospital, Angers
  - Nice University hospital, Nice

IPD SHARING:
Plan to Share IPD: No